CLINICAL TRIAL: NCT05589883
Title: Pilot Feasibility of the Cultural Adaptation of EMPOWER for Latinx Informal Caregivers in Intensive Care Units in the Context of COVID-19
Brief Title: A Study of the EMPOWER Program for Latinx Caregivers of ICU Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-141
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Informal Caregiver
Keywords: EMPOWER Program; Latinx Caregivers; ICU Patients; 22-141

STUDY DESIGN:
Intervention Model Description: The design of this study is a single-arm open trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMPOWER-Latinx intervention (Experimental): Informal caregivers will meet with the interventionist one-on-one via telepsychiatry (e.g., WebEx, Zoom) for 6, 15-20 minute modules to be completed within about 2-3 days from initiation of the first module, not including the booster modules. Informal caregivers will complete study assessments as per the schedule of assessments.
  Interventions: Behavioral: EMPOWER-Latinx

INTERVENTIONS:
Behavioral: EMPOWER-Latinx — EMPOWER-Latinx will be delivered in Spanish by videoconferencing (i.e., Zoom, WebEx) with a trained study interventionist. Intervention modules will be audio- and video-recorded (videorecording optional).

SUMMARY:
The researchers are doing this study to find out whether EMPOWER (Enhancing & Mobilizing the Potential for Wellness & Emotional Resilience) may reduce emotional distress in Latinx caregivers of patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers of patients, who were admitted in an ICU or step-down unit during their current admission/stay or within 2 weeks of discharge from their last admission/stay.
* Informal caregivers listed as a designated health care proxy or decision-making patient surrogate by ICU medical staff.
* Age 18 years or older as per self-report.
* Residing in New York or New Jersey as per self-report or able to complete modules while complying with current telehealth regulations.
* Spanish-speaking as per the Spanish language assessment items below and willing to receive the intervention in Spanish.

  * What is the participant's preferred language?
  * (Specify Lang)___________________________
  * How well does the participant speak Spanish?
  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)

Exclusion Criteria:

* Informal caregivers who score low, moderate or high on the Columbia Suicide Severity Rating Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
feasibility of EMPOWER-Latinx | 1 year
  Targets will include completion of 4/6 modules for feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Rosairo Costas Muniz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm